CLINICAL TRIAL: NCT00428857
Title: Noninvasive Ventilatory Support After Lung Surgery to Prevent Pulmonary Complications in COPD Patients
Brief Title: Noninvasive Ventilatory Support After Lung Surgery in COPD Patients
Acronym: POPVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P070501
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2007-01

CONDITIONS: COPD; Post Pulmonary Resection
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

INTERVENTIONS:
Procedure: non invasive ventilation — non invasive ventilation

SUMMARY:
Rationale: respiratory complications are the most frequent complications following lung resection and represent a noticeable cause of mortality. Benefits from non-invasive ventilation (NIV) in acute respiratory failure are now clearly demonstrated. The use of preventive NIV after lung resection, in the absence of acute respiratory failure and/or hypercarbia, could be justified by the physiological benefits expected. The goal of this study is to assess the efficacy of post-operative NIV in moderate-to-severe COPD, for prevention of respiratory complications.

Material and Methods: This is a prospective randomised multicenter trial with an open parallel design in moderate-t-o-severe COPD patients hospitalised in thoracic surgery for lung resection.

Expected results: This study will determine whether post-operative NIV decreases the incidence of acute respiratory events (acute respiratory failure) and whether some subgroups of patients benefit more from this strategy.

Conclusion: This study should help evaluating the utility of post-operative NIV after lung resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (FEV1 pre-operative <80% and FEV1/CV<70%)
* Patients undergoig pulmonary resection
* Informed consent

Exclusion Criteria:

* Apnea syndrom and chronic noninvasive support
* Post-operative extrarespiratory organ failure
* Inhability to follow study protocole
* Absence of medical coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: christine lorut, MD, Principal Investigator — APHP; antoine rabbat, MD, Principal Investigator — APHP
Locations (7):
- France (7):
  - Hopital Du Bocage, Dijon, Dijon
  - HEGP, Paris, Paris
  - hopital de Pontoise, Pontoise, Pontoise
  - CHU strasbourg, Strasbourg, Strasbourg
  - Hotel Dieu, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Larrey, Toulouse